CLINICAL TRIAL: NCT00917618
Title: The Effects of Group Cycling (Spinning®) On Gait and Pain-Related Disability in Persons With Knee Osteoarthritis: A Randomized Control Trial
Brief Title: The Effects of Group Cycling (Spinning®) With Knee Osteoarthritis: A Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Hospital, Pittsburgh, PA (Other)
Collaborators: PNC Band arthritis research fund (Unknown); Mad Dogg Athletics (Other)
Responsible Party: Sponsor
Organization: University of Pittsburgh (Other)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2009-06

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; knee; exercise; cycling
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise intervention (Active Comparator): Patients began the exercise intervention after randomization for 12 weeks
  Interventions: Other: Exercise
- Control (Placebo Comparator): Patients were asked not to change their baseline exercise program
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — Patients randomized to treatment arm attended 2-3 Spinning classes per week for 12 weeks.
  Arms: Exercise intervention
Other: Control — Patients randomized to the control arm were instructed not to change their baseline exercise programs
  Arms: Control

SUMMARY:
Hypothesis: Group cycling classes (Spinning®) will improve pain and functional outcomes in patients with knee osteoarthritis

Methods: Patients with symptomatic knee OA will be randomized to active Spinning® classes 2-3 per week or control group for 3 months. Outcomes including gait speed, WOMAC, KOOS, KOS, and VAS pain at rest and after 6 min walk will be performed at baseline and at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic and radiographic knee OA

Exclusion Criteria:

* severe patella femoral knee pain that would make cycling difficult
* medical condition which would prohibit an exercise program

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-01; Primary Completion 2006-05 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Preferred gait speed | 12 weeks

SECONDARY OUTCOMES:
WOMAC | 12 weeks
KOS | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Krohn, MD, Principal Investigator — Mercy Hospital of Pittsburgh
Locations (1):
- Mercy Hospital of Pittsbugh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Salacinski AJ, Krohn K, Lewis SF, Holland ML, Ireland K, Marchetti G. The effects of group cycling on gait and pain-related disability in individuals with mild-to-moderate knee osteoarthritis: a randomized controlled trial. J Orthop Sports Phys Ther. 2012 Dec;42(12):985-95. doi: 10.2519/jospt.2012.3813. Epub 2012 Aug 2. PMID 22951360